CLINICAL TRIAL: NCT03140241
Title: Pain Assessment by Pupil Dilation Reflex (PDR) and Pupillary Pain Index (PPI) in Response to Noxious Stimulation in Anesthetized Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, MD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/40/410-2
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Nociceptive Pain; Monitoring, Intraoperative
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDR measurement (Experimental): Two measurements of PDR perioperatively before and after opioid administration
  Interventions: Procedure: PDR measurement

INTERVENTIONS:
Procedure: PDR measurement — PDR measurement at two standardized times perioperatively:
  1. : anesthetized subject by propofol sedation until sedation depth monitor NeuroSense® (NeuroWave Systems Inc, Cleveland, OH) between 40-50
  2. : administration of remifentanil via effect site target concentration (Minto-model) at 5 ng/ml, in the absence of adjustments in sedation depth
  Other Names: PPI assessment

SUMMARY:
After conduction a pilot study, pupillary dilation reflex (PDR) is measured in response to nociceptive stimulation perioperatively.

DETAILED DESCRIPTION:
An infrared camera of the video pupillometer measures the pupillary dilation reflex (PDR) in response to incremental nociceptive stimuli. The PDR is a robust reflex, even in patients under general anesthesia, and may provide a potential evaluation of the autonomous nociceptive circuit. American Society of Anesthesiologists (ASA) classification I or II patients undergoing elective surgery under general anesthesia are recruited. Enrolled patients perioperative undergo PDR measurement at 2 different standardized times (before and after opioid administration) generated by an inbuilt pupillary pain index (PPI) protocol. PPI, as a surrogate for nociception includes noxious stimulations from 10 up to 60 milli ampere (mA) until pupil dilation is larger than 13% from baseline diameter. Therefore, no inappropriate high stimulation is executed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled abdominal or gynecological surgery
* ASA I-II

Exclusion Criteria:

* History of eye deformity, invasive ophthalmologic surgery
* Known cranial nerve(s) deficit
* Infection of the eye
* Predicted difficult airway management (DAF Guidelines)
* Chronic opioid use (>3 months)
* Ongoing treatment with beta-blockers, dopamine antagonists, topical atropine
* Preoperatively administrated benzodiazepins or antiemetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Stimulation Intensity | During perioperative period
  Necessary stimulation intensity to dilate the pupil more than 13%

SECONDARY OUTCOMES:
Pupillary Pain Index score | During perioperative period
  Device specific PPI score defined in accordance to stimulation intensity necessary for pupil dilation more than 13%
Systolic blood pressure | During PDR measurements
  Hypertension as a common used parameter for perioperative nociceptive assessment
Heart rate | During PDR measurements
  Tachycardia as a common used parameter for perioperative nociceptive assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Baeten, MD, Principal Investigator — University Hospital, Antwerp; Natasja Peeters, MD, Principal Investigator — University Hospital, Antwerp; Vera Saldien, MD, Study Chair — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication — https://www.ncbi.nlm.nih.gov/pubmed/29671874